CLINICAL TRIAL: NCT01158989
Title: Clinical Evaluation of Endoscopic Video Capsule for Investigation of Small Intestine Transit Time and Intestinal Pathology in Critically Ill Patients
Brief Title: Clinical Evaluation Gastrointestinal Motility With PillCam
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Responsible Party: Sponsor
Other Study IDs: PillCam
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Gastrointestinal Motility
Keywords: Critical care; Endoscopy, Video Capsule; Nutrition, Enteral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Critically ill: Critically ill subjects were intubated, mechanically ventilated and sedated
  Interventions: Device: PillCam
- Ambulatory Group: Subjects were scheduled for an outpatient procedure but were otherwise healthy
  Interventions: Device: PillCam

INTERVENTIONS:
Device: PillCam — Within four days of hospital admission, qualifying critically ill patients were assigned to the study and received a gastro-jejunal tube and one PillCam video telemetry capsule (Given Imaging Ltd., Yoqneam, Israel). In each critical care patient, placement of the video capsule was coupled with the placement of the medically necessary feeding tube. A flexible endoscope was inserted into the patient's mouth, and then advanced into the esophagus, stomach, and upper small intestine. The capsule was placed into a capsule delivery device and released into the distal duodenum after it had passed beyond the sight of the scope; a wire was placed to facilitate passage of the feeding tube. An abdominal X-ray was obtained to confirm feeding tube tip placement.
  Other Names: PillCam video telemetry capsule, Given Imaging Ltd.

SUMMARY:
The purpose of this study is to evaluate the clinical usefulness of a video camera pill (PillCam) in assessing intestinal function in the small intestines of patients. It is believed that the condition of the subjects digestive system can have a large impact on their overall physical health. Therefore, the investigators would like to assess whether using the pill device helps to determine any functional problems in patients in the ICU. The investigators are studying ICU patients because any change in their condition can have a large impact on their recovery. The same device will be used in healthy subjects scheduled for elective ambulatory surgery.

ELIGIBILITY:
Inclusion Criteria:

* mild-to-moderate brain injury patients who suffered from traumatic or non-traumatic intracranial hemorrhage
* admitted to an intensive care unit (ICU)
* needed an enteral tube placed for feeding
* control (ambulatory) group consisted of outpatients with no history of major abdominal surgery

Exclusion Criteria:

* younger than 18 years
* suffered multiple injuries (especially abdominal trauma or inflammatory bowel disease)
* had a history of complicated or unknown abdominal surgery
* presented with clinical evidence of ileus or suspected obstruction
* Patients with a pacemaker

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients (i.e., all were intubated, mechanically ventilated and sedated) and healthy patients scheduled for an outpatient procedure.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2006-05; Primary Completion 2007-11 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
small bowel transit times | 8 hours
  Small bowel transit time was calculated by measuring the difference between the start-time (i.e., placement of the capsule in the duodenum) and end-time (i.e., capsule enters the cecum). Examination of the differences between subsequent images indicates the amount of capsule movement and is proportional to the instant velocity ("motility") of the capsule

SECONDARY OUTCOMES:
visualization | 8 hours
  The quality of the visualization was determined using a three-step scale: Grade 0: intraluminal fluid disturbed visualization and significantly impaired interpretation: grade 1: intraluminal fluid present but did not impair visualization or interpretation; grade 2: no intraluminal fluid, excellent visualization

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Rauch, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Hospital, Louisville, Kentucky, United States